CLINICAL TRIAL: NCT02717338
Title: Blood Donor Competence, Autonomy and Relatedness Enhancement (Blood Donor CARE)
Brief Title: Blood Donor Competence, Autonomy and Relatedness Enhancement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: New York Blood Center (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Christopher R. France, Ph.D., Distinguished Professor, Ohio University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NHLBI R01HL127766; R01HL127766 (NIH)
Record Dates: First submitted 2016-02-18; First posted 2016-03-23 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Blood Donors
Keywords: blood donor; retention; motivation; self-determination theory
MeSH Terms: interventions — Mental Competency; Phylogeny

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Competence (Experimental): Participants will be assigned to review our donor coping website.
  Interventions: Behavioral: Competence
- Autonomy (Experimental): Participants will be assigned to receive a brief telephone interview.
  Interventions: Behavioral: Autonomy
- Relatedness (Experimental): Participants will be asked to join a closed Facebook group for one month.
  Interventions: Behavioral: Relatedness
- Competence + Autonomy (Experimental): Participants will be assigned to the web site review, followed by the brief telephone interview.
  Interventions: Behavioral: Competence; Behavioral: Autonomy
- Competence + Relatedness (Experimental): Participants will be assigned to the web site review, followed by the one-month Facebook group membership.
  Interventions: Behavioral: Competence; Behavioral: Relatedness
- Autonomy + Relatedness (Experimental): Participants will be assigned to the brief telephone interview, followed by the one-month Facebook group membership.
  Interventions: Behavioral: Autonomy; Behavioral: Relatedness
- Competence + Autonomy + Relatedness (Experimental): Participants will be assigned to the web site review, brief telephone interview, and one-month Facebook group membership.
  Interventions: Behavioral: Competence; Behavioral: Autonomy; Behavioral: Relatedness
- Treatment-as-Usual Control (No Intervention): Participants will receive the standard communications that New York Blood Center has with all first-time donors.

INTERVENTIONS:
Behavioral: Competence — Participants will be assigned to review our donor coping website that combines text, videos, and interactive features to directly address common donor fears and to offer advice on empirically-validated strategies to reduce fear, pain, and syncopal reactions.
  Arms: Competence; Competence + Autonomy; Competence + Autonomy + Relatedness; Competence + Relatedness
Behavioral: Autonomy — Participants will be assigned to receive a brief telephone interview that we have developed that encourages blood donors to reflect upon their unique motivations for giving and how the act of donating is consistent with their broader life goals and values.
  Arms: Autonomy; Autonomy + Relatedness; Competence + Autonomy; Competence + Autonomy + Relatedness
Behavioral: Relatedness — Participants will be asked to join a closed Facebook group for one month. The group encourages participants to discuss their experiences with blood donation, including such things as posting images of their donations and/or reasons for donating. Posts will be designed to encourage social interaction around donation experiences, identity formation and group affiliation.
  Arms: Autonomy + Relatedness; Competence + Autonomy + Relatedness; Competence + Relatedness; Relatedness

SUMMARY:
The purpose of this study is to determine whether enhancing blood donor competence, autonomy, and/or relatedness increases intrinsic motivation to donate and improves donor retention.

DETAILED DESCRIPTION:
For health, safety, and economic reasons there is a critical need for novel approaches to enhance the retention of new blood donors. The current study examines an innovative, theory-driven approach to retention by promoting intrinsic motivation to donate again among new blood donors. Self-determination theory (SDT) proposes that people are more likely to persist with behaviors that are internally versus externally motivated, and considerable research supports the notion that more internalized motivation is associated with better adherence in a variety of health contexts. Similar findings have also been reported in the blood donation context where measures of the extent to which a donor identity has been internalized are positively related to both donation intention and future donation behavior. Based on prior work, the investigators propose to test a multi-component intervention designed to enhance one, two, or all three of the fundamental human needs that contribute to internal motivation according to SDT (i.e., competence, autonomy, relatedness). Using a full factorial design, first-time donors will be randomly assigned to a control condition or an intervention that addresses one, two, or all three of the fundamental needs. The primary aim is to determine whether the intervention conditions, alone and in combination, increase the likelihood of a donation attempt in the next year. The second aim is to examine intervention-specific increases in competence, autonomy, and relatedness as potential mediators of enhanced donor retention. Finally, an exploratory aim will examine an integrative model of motivation that views autonomy as a mediating influence on the more proximal, situational-level determinants of behavior (i.e., attitude, subjective norm, perceived behavioral control, and intention).

ELIGIBILITY:
Inclusion Criteria:

* First-time whole blood donor with New York Blood Center;
* Eligible to donate again;
* Willing to be randomly assigned;
* Have, or be willing to establish, an active Facebook account.

Exclusion Criteria:

* History of more than one lifetime whole blood donation (with any blood center);
* Ineligible to donate again (based on New York Blood Center donor eligibility determination);
* Unwilling to be randomly assigned;
* Unwilling to sign up for closed Facebook group, if randomly assigned.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2580 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Repeat Blood Donation Attempts | one year plus 8 weeks post-initial donation
  Donor records will be used to track all instances of subsequent donation attempts during the one-year follow-up.

SECONDARY OUTCOMES:
Blood Donation Attitude | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Subjective Norms | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Perceived Behavioral Control | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Intention | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Personal Moral Norm | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Anticipated Regret | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Donation Anxiety | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Decisional Balance Inventory for Blood Donation | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donation Ambivalence Scale | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donor Identity Survey | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donor Action and Coping Self-Efficacy | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Blood Donor Relatedness Scale | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Social Media Use Scale | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.
Social Media Relatedness Scale | Pre-intervention (requested 1-2 weeks post-donation) and Post-intervention (requested 7 weeks post-donation)
  Participant receives email request to complete online questionnaire at specified times.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. France, Ph.D., Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Following publication of our findings, the raw and processed data will be freely available to any researcher who requests a copy. The raw data files will be stored as EXCEL and SPSS data files and will be de-identified so there is no possibility of connecting the information with the original participants. To obtain access to the data, interested parties can contact the PI.
Supporting Information: Study Protocol, ICF
Time Frame: De-identified data will be made available one year after publication of the study findings.
Access Criteria: A controlled access approach will be used to share de-identified data with individuals who 1) make an official request to the Principal Investigator, 2) demonstrate a legitimate academic purpose for the request, 3) provide evidence of up-to-date compliance with human subjects ethics training, and 4) agree to delete the data within an agreed-upon timeframe and not share the data with others.

REFERENCES:
- [Result] France CR, France JL, Himawan LK, Fox KR, Livitz IE, Ankawi B, Slepian PM, Kowalsky JM, Duffy L, Kessler DA, Rebosa M, Rehmani S, Frye V, Shaz BH. Results from the blood donor competence, autonomy, and relatedness enhancement (blood donor CARE) randomized trial. Transfusion. 2021 Sep;61(9):2637-2649. doi: 10.1111/trf.16577. Epub 2021 Jul 5. PMID 34224590
- [Derived] Frye V, Duffy L, France JL, Kessler DA, Rebosa M, Shaz BH, Carlson BW, France CR. The Development of a Social Networking-Based Relatedness Intervention Among Young, First-Time Blood Donors: Pilot Study. JMIR Public Health Surveill. 2018 Apr 26;4(2):e44. doi: 10.2196/publichealth.8972. PMID 29699961
- [Derived] France CR, France JL, Carlson BW, Frye V, Duffy L, Kessler DA, Rebosa M, Shaz BH. Applying self-determination theory to the blood donation context: The blood donor competence, autonomy, and relatedness enhancement (Blood Donor CARE) trial. Contemp Clin Trials. 2017 Feb;53:44-51. doi: 10.1016/j.cct.2016.12.010. Epub 2016 Dec 12. PMID 27979752

DOCUMENTS (3):
  • Informed Consent Form: Adult Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02717338/ICF_000.pdf
  • Informed Consent Form: Child Assent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02717338/ICF_001.pdf
  • Informed Consent Form: Parental Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/38/NCT02717338/ICF_002.pdf